CLINICAL TRIAL: NCT02392455
Title: Vargatef in 2nd-line Therapy of Advanced or Metastatic Adenocarcinoma of the Lung
Brief Title: VARGADO - Vargatef in 2nd-line Therapy of Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199.211; 1199-0211 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2015-03-17; First posted 2015-03-19 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- A
  Interventions: Drug: treatment

INTERVENTIONS:
Drug: treatment — Docetaxel plus nintedanib until progression or intolerability

SUMMARY:
This observational study will investigate the efficacy and tolerability of Vargatef (Nintedanib) plus docetaxel in daily routine second-line treatment in patients with locally advanced, metastatic or locally recurrent NSCLC. Treatment with Vargatef in eligible NSCLC patients, for whom the treating physician has decided to initiate treatment with Vargatef in second line according to the local label, will be observed for up to 24 months. Survial follow-up will be done until the end of the study.

ELIGIBILITY:
Inclusion criteria:

* age 18 or older
* men and women locally advanced, metastastic and/or recurrent NSCLC with adenocarcinoma histology for which vargatef treatment is indicated according to Summary of Product Characteristics (SmPC)
* after first line chemotherapy. This includes also combinations of immune- and chemotherapy.
* standard 21-day-cycles docetaxel treatment according to SmPC possible
* written informed consent

Exclusion criteria:

* contraindications according to the SmPC of Vargatef or Docetaxel
* more than one chemotherapy for treatment of NSCLC in palliative setting
* current partcipation in a clinical trial
* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients
Sampling Method: Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Percentage of patients alive one year after start of therapy with Vargatef and Docetaxel (1-year survival rate) | up to 24 months

SECONDARY OUTCOMES:
One year survival rate of patients with first line progression within 9 months after start of first line therapy | up to 24 months
Progression-free survival of patients with first line progression within 9 months after start of first line therapy | up to 24 months
Median overall survival | up to 24 months
Progression-free survival | up to 24 months
Tumour control rate (complete response, partial response, stable disease) | up to 24 months
Incidence of side effects | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Grohe C, Blau W, Gleiber W, Haas S, Hammerschmidt S, Kruger S, Muller-Huesmann H, Schulze M, Wehler T, Atz J, Kaiser R. Real-World Efficacy of Nintedanib Plus Docetaxel After Progression on Immune Checkpoint Inhibitors: Results From the Ongoing, Non-interventional VARGADO Study. Clin Oncol (R Coll Radiol). 2022 Jul;34(7):459-468. doi: 10.1016/j.clon.2021.12.010. Epub 2022 Jan 7. PMID 35012901
- [Derived] Grohe C, Gleiber W, Haas S, Losem C, Mueller-Huesmann H, Schulze M, Franke C, Basara N, Atz J, Kaiser R. Nintedanib plus docetaxel after progression on immune checkpoint inhibitor therapy: insights from VARGADO, a prospective study in patients with lung adenocarcinoma. Future Oncol. 2019 Aug;15(23):2699-2706. doi: 10.2217/fon-2019-0262. Epub 2019 Jul 8. PMID 31282758
- See also: Related Info — https://www.mystudywindow.com